CLINICAL TRIAL: NCT07081516
Title: The Effect of Intrathecal Bupivacaine Temperature Variation on Prophylaxis of Post-Spinal Shivering in Urologic Patients Undergoing Spinal Anesthesia (A Randomized, Controlled, Double-Blinded Study)
Brief Title: Effect of Intrathecal Bupivacaine Temperature Variation on Prophylaxis of Shivering in Urologic Patients Undergoing Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Emad Mohamed Ahmed Abdelhafez, Lecturer of Anesthesia, Critical Care and Pain Management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-4-2025
Record Dates: First submitted 2025-07-08; First posted 2025-07-23 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Shivering, Spinal Anesthesia
MeSH Terms: interventions — Temperature

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (cold group)patients will be given 15 mg Bupivacaine 0.5% plus Fentanyl 25 ug at (4°C) temp (Active Comparator)
  Interventions: Procedure: temperature
- Group B (Room temp group) patients given 15 mg Bupivacaine 0.5% plus Fentanyl 25 ug at (24°C) temp (Active Comparator)
  Interventions: Procedure: temperature
- Group C (Warm group) patients given15 mg Bupivacaine 0.5% plus Fentanyl 25 ug at (37 °C) temp (Active Comparator)
  Interventions: Procedure: temperature

INTERVENTIONS:
Procedure: temperature — Adjusting the temperature of the local anesthetic drugs injected intrathecally

SUMMARY:
The aim of this study is to evaluate the effect of temperature variation of injected intrathecal bupivacaine on prophylaxis of post-spinal shivering in urological patients undergoing spinal anaesthesia.

DETAILED DESCRIPTION:
Preoperative:

After obtaining informed consent the day before surgery by an anesthetist who is not involved in the study from the patient. Subjects with contraindications to regional anaesthesia will be excluded. A history will be taken from all patients. Age and American Society Anesthesiologists' (ASA) score will be recorded. Laboratory investigations including complete blood picture, coagulation profile, liver and renal functions will be recorded. General examination will be conducted with examination of the back to exclude infection at the injection site and anatomical deformities.

Intra-operative:

The study consists of three groups: group A, group B and group C

* Group A patients will be injected with 15 mg heavy bupivacaine 0.5% (equals to a volume of 3 ml) intrathecally plus 25 µg fentanyl that is adjusted to temperature of (4°C) by being stored in a pharmaceutical refrigerator by adjusting its thermostat to be on 4°C and consists of 18 patient.
* Group B patients will be injected with 15 mg heavy bubivacaine 0.5% (equals to a volume of 3 ml) intrathecally plus 25 µg fentanyl that is stored at room temperature of (24°C) by adjusting the temperature settings of the air conditioning and consists of 18 patient.
* Group C patients will be injected with 15 mg heavy bupivacaine 0.5% (equals to a volume of 3 ml) intrathecally plus 25 µg fentanyl that is adjusted to temperature of (37 °C) by using a fluid warming cabinet adjusted to be on 37 °C and consists of 18 patients.

Upon arrival to the operation room; perioperative monitoring will include continuous Electrocardiogram, pulse oximetry, non-invasive arterial blood pressure measurement and temperature measurement, baseline vital signs will be recorded and an IV access will be secured.

To facilitate blinding, a two operator technique will be employed. The study drugs will be prepared by an investigator who is not involved in patient handling.

The drugs will be prepared according to the group selected by the closed envelope method in syringes coded to the group, patient name and number.

Strict aseptic technique is necessary, it will be achievable with adequate hand-washing, mask and cap use, and chlorhexidine antiseptics with alcohol content, Cleaning of the site of injection always starts from the chosen site of approach in circles and then away from the site. Time will be allowed for the cleaning solution to dry then Local anesthetic (about 1 mL of 2% lidocaine) is used for skin infiltration, and a wheal is created at the site of access chosen.

Spinal anesthesia will be performed in the sitting position at the L4-L5 interspace with a midline approach, using a 25-gauge Quincke needle by an anesthetist who is blind to the temperature of the drugs injected then the patient will be placed in the supine position. All intravenous fluids infused will be warmed up to 37 °C and all patients will be covered by a single standard blanket that is not actively warmed.

Sensory anesthesia will evaluated by a second anaesthetist unaware at which temperature the drug was injected using pinprick test to confirm a blockade at T10 dermatome or more and onset of motor blockade will be evaluated by asking the patient to flex their knees and ankles.

Blood pressure will be recorded at intervals of 5 min. for the first 30 minutes and every 15 min. for the rest of operation time.

The primary outcome is the incidence of shivering during the whole observation period from the time of the block till the patient is discharged from the post anaesthesia care unit as defined by shivering score (12) ≥ 3. The shivering score will be assessed at 10min intervals after the spinal block and graded by the four-point scale validated by Wrench et al.

Grade 0: No Shivering. Grade 1: One or more of the following: Piloerection, peripheral vasoconstriction, peripheral cyanosis, but without visible muscle activity Grade 2: Visible muscle activity confined to one muscle group Grade 3: Visible muscle activity in more than 1 muscle group Grade 4: Gross muscle activity involving the whole body. Shivering grade ≥ 3 will be recorded once it happens as a yes or no. The patients will be recorded for the start of shivering after spinal anesthesia (onset of shivering), severity of shivering (its grade), time of disappearance (duration of shivering) and response rate (shivering ceasing within 15 min after treatment).

Non pharmacological measures like covering the patient with a warm blanket and providing verbal reassurance can help reduce anxiety, which can sometimes contribute to shivering. Continuous shivering of grade 3 or 4 for more 15 min will be treated with pethidine (0.5 mg/kg IV) and Patients who did not respond or in whom recurrence of shivering occurred were treated with additional dose of pethidine (0.25 mg/kg IV).

Other adverse effects in the form of hypotension (mean arterial blood pressure < 20% of the baseline) will be treated with ephedrine 5-10 mg IV, bradycardia (< 50/ min) will be treated with atropine 0.5 mg IV, Pruritus will be treated with diphenhydramine 25 mg IV. Nausea and vomiting will be recorded as yes or no and ondasterone 4 mg IV will be administered for moderate to severe nausea and vomiting.

Tympanic temperature in Celsius (°C) will be recorded every 20 minutes and room temperature will be maintained at 24°C by adjusting the temperature settings of the air conditioning.

Duration of surgery will be noted and recorded

Post-operative:

In the post anaesthesia care unit, the motor blockade will be assessed with the Bromage scale (13) (1, unable to move feet; 2, able to move feet only; 3, just able to move the knees; and 4, full flexion of knees and feet).

Post-operative pain will be assessed according to VAS (14) (visual analogue scale) by the second anesthetist who is blinded to study group. Patient will be asked to rate average pain they experience over 24 hours post operatively on a 10 cm VAS: no pain - 0, very severe pain - 10. If VAS >3, the patient will receive analgesia in the form of nalbuphine 0.1 mg/kg maximum single dose 20 mg. maximum daily dose does not exceed 160 mg.

All patients will be followed up on the first and second postoperative days regarding occurrence of post puncture headache, backache, paresthesia, or hematoma at the site of injection.

The investigators who will collect and analyze the data will be blind to the group allocation and all patients and care givers will be unaware of the administered study drugs.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients scheduled for urological procedures under spinal anaesthesia. 2. Patient age ranges from 18 to 60 years. 3. American Society of Anesthesiologists (ASA) physical status class I or II.

Exclusion Criteria:

* 1. Patient's refusal of regional block. 2. Patients with neurological disorders, increased intracranial pressure, convulsive disorders, autonomic neuropathies, psychological disorders, or those lacking cooperation.

  3. Patients with anatomical abnormalities, skin lesions, wounds, or infection at the site of injection, or general infection.

  4. Patients with bleeding disorders defined as (INR>1.4) and/or (platelet count < 100,000/µL).

  5. Patients with known hypersensitivity to any of the study drugs. 6. Patients with renal impairment. 7. Patients with hepatic disease e.g. severe liver cell failure, or hepatic malignancy, or hepatic enlargement.

  8. Patients with failed, or partial spinal block.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Shivering | starting from the time of the spinal injection (T0) till the discharge from the PACU
  the incidence of grade 3 or 4 shivering which will be assessed at 10min intervals starting from the time of spinal block (T0) till the discharge from PACU. and it will be graded according to Wrench scale for shivering.
  Grade 0: No Shivering. Grade 1: One or more of the following: Piloerection, peripheral vasoconstriction, peripheral cyanosis, but without visible muscle activity Grade 2: Visible muscle activity confined to one muscle group Grade 3: Visible muscle activity in more than 1 muscle group Grade 4: Gross muscle activity involving the whole body.

CONTACTS AND LOCATIONS:
Overall Officials: Emad Mohamed Emad M. Abdelhafez00, Lecturer, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy Hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No